CLINICAL TRIAL: NCT02498392
Title: A Phase 2a Randomized, Double-blind, Placebo-Controlled, Parallel-Group, Multi-center Study Investigating the Efficacy, Safety, and Tolerability of JNJ-42165279 in Subjects With Major Depressive Disorder With Anxious Distress
Brief Title: An Efficacy, Safety and Tolerability Study of JNJ-42165279 in Participants With Major Depressive Disorder With Anxious Distress
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR107733; 2015-002007-29 (EudraCT Number); 42165279MDD2001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2015-07-13; First posted 2015-07-15 (Estimated); Results first posted 2022-04-07 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Depressive Disorder; Anxiety
Keywords: Major Depressive Disorder; Depression; Anxiety symptoms; JNJ-42165279
MeSH Terms: conditions — Depressive Disorder; Anxiety Disorders; Depressive Disorder, Major; Depression | interventions — JNJ-42165279

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (4):
- Responders-Placebo (Placebo Comparator): Participants who responded in the placebo lead-in period will be administered with Matching Placebo orally.
  Interventions: Other: Placebo
- Responders-JNJ-42165279 (Experimental): Participants who responded in the placebo lead-in period will be administered with JNJ-42165279 orally at a dose of 25 milligrams (mg) tablets once daily for 6 weeks.
  Interventions: Drug: JNJ-42165279
- Non Responders-Placebo (Placebo Comparator): Participants who did not respond in the placebo lead-in period will be administered with Matching Placebo orally.
  Interventions: Other: Placebo
- Non Responders-JNJ-42165279 (Experimental): Participants who did not respond in the placebo lead-in period will be administered with JNJ-42165279 orally at a dose of 25 mg tablets once daily for 6 weeks.
  Interventions: Drug: JNJ-42165279

INTERVENTIONS:
Drug: JNJ-42165279 — JNJ-42165279 will be administered orally at a dose of 25 milligrams (mg) tablet once daily for 6 weeks.
  Arms: Non Responders-JNJ-42165279; Responders-JNJ-42165279
Other: Placebo — Matching Placebo will be administered orally.
  Arms: Non Responders-Placebo; Responders-Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety and tolerability of JNJ-42165279 in participants with major depressive disorder (MDD) with anxiety symptoms who have had inadequate response to treatment with a selective serotonin reuptake inhibitor (SSRI) or serotonergic/noradrenergic reuptake inhibitor (SNRI).

DETAILED DESCRIPTION:
This is a multicenter, double-blind (neither physician nor participant knows the treatment that the participant receives), placebo-controlled, randomized, parallel-group study in participants with Major Depressive Disorder (MDD) with Anxious Distress. Participants who had treatment initiated with a SSRI/SNRI allowed by the protocol will be evaluated at the investigation site. The site assessment will be reviewed and validated by an independent central rater. The review will include the clinical history of MDD, SSRI/SNRI treatment of adequate dose and duration for the current episode of depression, and current symptom severity on the Hamilton Depression Rating Scale (HDRS17). Enrolled participants will be maintained on SSRI/SNRI treatment throughout the study to determine whether additional treatment with JNJ-4216579 can reduce the symptoms of MDD with anxious distress.The study will consist of 3 phases: a Screening Phase of up to 4 weeks, an 11-week double-blind Treatment Phase, and a 3-week post-treatment (follow up) Phase. The double-blind treatment Phase of the trial will consist of 3 periods. The first period is a placebo lead-in of double-blind duration, after which participants will enter the treatment period when they will be randomly assigned to JNJ-42165279 or continuation on placebo for 6 weeks. Participants who successfully complete the treatment period prior to the end of Week 11, will be treated with placebo for the remaining time of the double-blind phase of the study, which will vary depending on the duration of the placebo lead-in for the specific participant. The total study duration for each participant will be approximately 18 weeks. Efficacy and safety of JNJ-42165279 will be evaluated. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant must meet the Diagnostic and Statistical Manual of Mental Disorders-IV (DSM-IV) or 5 diagnostic criteria for major depressive disorder (MDD) with Anxious Distress
* Participants with a diagnosis of comorbid Generalized Anxiety Disorder, Social Anxiety Disorder, or Panic Disorder may be included, if the investigator considers MDD with Anxious Distress to be the primary diagnosis (confirmed by an independent central rater at screening)
* Participants must have been treated with an approved SSRI/SNRI antidepressants for at least 6 continuous weeks, validated by an independent central rater contracted by the sponsor
* A 17-item Hamilton Depression Rating Scale (HDRS17) total score greater than or equal to (>=)18 and a HDRS17 anxiety/somatization factor score >=7 at screening, assessed by a site rater and reviewed by an independent central rater on Day 1
* Participant must be willing and able to adhere to the prohibitions and restrictions
* Participant Body mass index (BMI = weight/height2) must be between 18 and 35 kilogram per square meter (kg/m^2) inclusive

Exclusion Criteria:

* Has other psychiatric condition, including, but not limited to, MDD with psychotic features, bipolar disorder, obsessive-compulsive disorder, post-traumatic stress disorder, borderline personality disorder, eating disorder, or schizophrenia
* Has a length of current Major Depressive Episode (MDE) greater than (>) 6 months
* Has more than 1 failed antidepressant treatment of adequate dose and duration in the current MDE, Not including the inadequate response to the current selective serotonin reuptake inhibitor (SSRI) or serotonergic/noradrenergic reuptake inhibitor (SNRI) antidepressant
* Has initiated psychotherapy specific for MDD (such as cognitive behavioral, behavioral, or interpersonal therapy) for the current episode of depression within 6 weeks prior to Screening
* Has a current or recent history of clinically significant suicidal ideation within the past 6 months, or a history of suicidal behavior within the past year

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 161 (Actual)
Dates: Start 2015-10-07 (Actual); Primary Completion 2019-02-04 (Actual); Study Completion 2019-02-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (32):
- United States (8):
  - Costa Mesa, California
  - Oceanside, California
  - Miami, Florida
  - Natick, Massachusetts
  - Cedarhurst, New York
  - Raleigh, North Carolina
  - Allentown, Pennsylvania
  - Salt Lake City, Utah
- Chisinau, Moldova
- Russia (5):
  - Orenburg
  - Saint Petersburg
  - Saratov
  - Tomsk
  - Yekaterinburg
- Spain (5):
  - Alicante
  - Barcelona
  - Bilbao
  - Sant Boi de Llobregat
  - Zamora
- Ukraine (7):
  - Hlevakha
  - Kharkiv
  - Kherson
  - Kyiv
  - Lviv
  - Smila
  - Uzhhorod
- United Kingdom (6):
  - Barnsley
  - Blackpool
  - Liverpool
  - Manchester
  - South Staffordshire
  - Stourton

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 161 enrolled participants, 1 participant withdrew from study participation prior to dosing. This participant has not been included in the analysis.
Groups:
- Placebo: All participants received matching placebo tablets orally once daily (qd) during the double blind lead-in period. Participants were then assessed for response according to criteria based on reduction from lead-in baseline in Hamilton depression rating scale (HDRS17) and continued to receive adjunctive matching placebo tablets orally qd for 6 weeks during the double-blind treatment period. Participants who completed the double-blind treatment period prior to Week 11 entered the withdrawal period and were treated with placebo for the remaining time of the treatment phase of the study, which varied depending on the duration of the placebo lead-in for the specific participant.
- JNJ-42165279 25 mg: Participants receiving matching placebo tablets during the double blind lead-in period were randomized to receive JNJ-42165279 25 milligrams (mg) tablets orally qd for 6 weeks during the double-blind treatment period. Participants who completed the double-blind treatment period prior to Week 11 entered the withdrawal period and were treated with placebo for the remaining time of the treatment phase of the study, which varied depending on the duration of the placebo lead-in for the specific participant.
Period: Double-blind(DB) Lead-in Period(3 Weeks)
Arm/Group | Placebo | JNJ-42165279 25 mg
Started | 160 | 0
Treated | 153 | 0
Completed | 153 | 0
Not Completed | 7 | 0
Not completed — Did not receive treatment | 7 | 0
Period: DB Treatment (6 Weeks)+Withdrawal Period
Arm/Group | Placebo | JNJ-42165279 25 mg
Started | 76 | 77
Completed | 70 | 67
Not Completed | 6 | 10
Not completed — Adverse Event | 3 | 0
Not completed — Lack of Efficacy | 0 | 2
Not completed — Lost to Follow-up | 0 | 2
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Other | 1 | 3

BASELINE CHARACTERISTICS:
Population: Baseline population is based on safety analysis set which included all enrolled participants who received at least one dose of study medication in the Lead-in Period and who were lead-in placebo non-responders.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | JNJ-42165279 25 mg | Total
Number analyzed (Participants) | 76 | 77 | 153
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.4 (11.92) | 42.1 (11.96) | 43.2 (11.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 53 | 112
  Male | 17 | 24 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 6 | 13
  Not Hispanic or Latino | 67 | 71 | 138
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 3 | 3
  White | 73 | 72 | 145
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  MOLDOVA, REPUBLIC OF | 8 | 10 | 18
  RUSSIAN FEDERATION | 20 | 21 | 41
  SPAIN | 3 | 3 | 6
  UKRAINE | 18 | 18 | 36
  UNITED KINGDOM | 18 | 17 | 35
  UNITED STATES | 9 | 8 | 17

OUTCOME MEASURES:

1. Primary Outcome: Double-blind Treatment Period: Change From Baseline in Hamilton Depression Rating Scale (HDRS17) Total Score at Week 6 (eITT Population)
Description: HDRS17 is clinician-administered rating scale designed to assess severity of symptoms in participants diagnosed with depression. Each of 17 items is rated by clinician on either 3-point (0-2) or 5-point (0-4) scale with rating of 0: absent, 1: doubtful to mild, 2: mild to moderate, 3: moderate to severe, and 4: very severe. A total score (0 to 52) was calculated by adding scores of all 17 items. For each item as well as total score, higher score represents more severe condition.
Time Frame: Baseline and Week 6
Population: The enriched intent-to-treat (eITT) analysis set included all enrolled participants who were randomized into double-blind treatment period, who were lead-in placebo non-responder, who received at least one dose of double-blind study medication (either placebo or JNJ-42165279) and had at least one post-baseline HDRS17 assessment in double-blind treatment period. Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | JNJ-42165279 25 mg
Number analyzed (Participants) | 47 | 47
Units on a scale | -6.1 (5.90) [lower limit 5.90] | -6.5 (4.01) [lower limit 4.01]
Statistical Analysis 1: Comparison: Placebo vs JNJ-42165279 25 mg; Test type: Superiority; p = 0.416, Mixed-effects Model for Repeated Measure; Difference of Least Square (LS) Means = -0.2, 60% CI 2-sided [-1.10 to 0.66], Standard Error of Mean 1.04

2. Primary Outcome: Double-blind Treatment Period: Change From Baseline in HDRS17 Total Score at Week 6 (fITT Population)
Description: HDRS17 is a clinician-administered rating scale designed to assess severity of symptoms in participants diagnosed with depression. Each of the 17 items is rated by clinician on either a 3-point (0 to 2) or a 5-point (0 to 4) scale which used a rating of 0: absent, 1: doubtful to mild, 2: mild to moderate, 3: moderate to severe, and 4: very severe. HDRS17 total score is calculated as sum of 17 item scores and ranges from 0 to 52. For each item as well as the total score, higher scores indicate greater severity of depression.
Time Frame: Baseline and Week 6
Population: The full intent-to-treat (fITT) analysis set included both placebo responders and placebo non-responders and defined as all enrolled participants who were randomized into the double-blind treatment period, who received at least one dose of double-blind study medication and had at least one post-baseline HDRS17 assessment during the double-blind treatment period. Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | JNJ-42165279 25 mg
Number analyzed (Participants) | 72 | 69
Units on a scale | -5.0 (6.34) [lower limit 6.34] | -5.2 (4.68) [lower limit 4.68]
Statistical Analysis 1: Comparison: Placebo vs JNJ-42165279 25 mg; Test type: Superiority; p = 0.647, Mixed-effects Model for Repeated Measure — 1-sided; Difference of Least Square (LS) Means = 0.3, 60% CI 2-sided [-0.41 to 1.07], Standard Error of Mean 0.88

3. Secondary Outcome: Double-blind Treatment Period: Change From Baseline in Hamilton Anxiety Rating Subscale (HAM-A6) Score at Week 6 (eITT Population)
Description: The HAM-A6 is a 6-item subscale derived from the original Hamilton Anxiety scale (HAM-A) which consists of 5 psychic anxiety symptoms (anxious mood, psychic tension, fears, intellectual disturbances, and anxious behavior observed at the interview), as well as one somatic item (muscular tension). Each of the 6 items is rated by the clinician on a 5-point scale ranging from 0 (not present) to 4 (maximum degree). The HAM-A6 score was calculated by summing the 6 item scores, and ranges from 0 to 24. Higher scores indicated greater severity of symptoms.
Time Frame: Baseline and Week 6
Population: The eITT analysis set included all enrolled participants who were randomized into double-blind treatment period, who were lead-in placebo non-responder, who received at least one dose of double-blind study medication (either placebo or JNJ-42165279) and had at least one post-baseline HDRS17 assessment in the double-blind treatment period. Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | JNJ-42165279 25 mg
Number analyzed (Participants) | 47 | 47
Units on a scale | -2.4 (3.15) [lower limit 3.15] | -2.9 (2.47) [lower limit 2.47]

4. Secondary Outcome: Double-blind Treatment Period: Change From Baseline in HAM-A6 Score at Week 6 (fITT Population)
Description: as for outcome 3
Time Frame: Baseline and Week 6
Population: The Full ITT (fITT) Analysis Set is defined as all enrolled participants who were randomized into the double-blind treatment period, who received at least one dose of double-blind study medication and have at least one post-baseline HDRS17 assessment during the double-blind treatment period. Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | JNJ-42165279 25 mg
Number analyzed (Participants) | 72 | 69
Units on a scale | -2.1 (3.12) | -2.2 (2.68)

5. Secondary Outcome: Double-blind Treatment Period: Change From Baseline in Hamilton Depression Rating Subscale (HAM-D6) Score at Week 6 (eITT Population)
Description: HAM-D6 is a 6-item subscale derived from HDRS17 and consists of depressed mood, guilt feelings, work and interests, psychomotor retardation, psychic anxiety, and somatics symptoms (tiredness and pain), rated on a 5-point scale, where 0 = not present, and 1-4 represent increasingly severe symptoms. Each of these items is rated by the clinician on either a 3-point (0 to 2) or a 5-point scale (0 to 4). The point scale used a rating of 0 (absent), 1 (doubtful to mild), 2 (mild to moderate), 3 (moderate to severe), and 4 (very severe). General somatic is scored 0 to 2 and all others are scored 0 to 4. The HAM-D6 is calculated from summing the 6 items and the score ranges from 0 (normal) to 22 (severe), with higher scores indicating greater severity of core symptoms.
Time Frame: Baseline and Week 6
Population: The eITT analysis set included all enrolled participants who were randomized into double-blind treatment period, who were lead-in placebo non-responder, who received at least one dose of double-blind study medication (either placebo or JNJ-42165279) and had at least one post-baseline HDRS17 assessment in double-blind treatment period. Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | JNJ-42165279 25 mg
Number analyzed (Participants) | 47 | 47
Units on a scale | -3.1 (3.20) [lower limit 3.20] | -3.6 (2.41) [lower limit 2.41]

6. Secondary Outcome: Double-blind Treatment Period: Change From Baseline in HAM-D6 Score at Week 6 (fITT Population)
Description: HAM-D6 is a 6-item subscale derived from HDRS17 and consists of depressed mood, guilt feelings, work and interests, psychomotor retardation, psychic anxiety, and somatic symptoms (tiredness and pain), rated on a 5-point scale, where 0 = not present, and 1-4 represent increasingly severe symptoms. Each of these items is rated by the clinician on either a 3-point (0 to 2) or a 5-point scale (0 to 4). The point scale used a rating of 0 (absent), 1 (doubtful to mild), 2 (mild to moderate), 3 (moderate to severe), and 4 (very severe). General somatic is scored 0 to 2 and all others are scored 0 to 4. The HAM-D6 is calculated from summing the 6 items and the score ranges from 0 (normal) to 22 (severe), with higher scores indicating greater severity of core symptoms.
Time Frame: Baseline and Week 6
Population: The fITT Analysis Set is defined as all enrolled participants who were randomized into the double-blind treatment period, who received at least one dose of double-blind study medication and have at least one post-baseline HDRS17 assessment during the double-blind treatment period. Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Unit on a Scale
Arm/Group | Placebo | JNJ-42165279 25 mg
Number analyzed (Participants) | 72 | 69
Unit on a Scale | -2.6 (3.30) | -2.8 (2.78)

7. Secondary Outcome: Double-blind Treatment Period: Change From Baseline in Structured Interview Guide of the Hamilton Anxiety Scale (SIGH-A) Total Score at Week 6 (eITT Population)
Description: The SIGH-A was included as a means to determine the frequency and severity of signs and symptoms of anxiety; and determine both their influence on treatment and their responsiveness to treatment. The SIGH-A scale consists of 14 items with a score of 0 to 4, where 0=absent, 1=mild, 2=moderate, 3=severe, 4=incapacitating. The SIGH-A total score is calculated by summing the 14 item scores, and ranges from 0 to 56. For each individual item score and total score, higher scores indicate greater severity.
Time Frame: Baseline and Week 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | JNJ-42165279 25 mg
Number analyzed (Participants) | 47 | 47
Units on a scale | -5.7 (7.11) [lower limit 7.11] | -6.8 (5.62) [lower limit 5.62]

8. Secondary Outcome: Double-blind Treatment Period: Change From Baseline in SIGH-A Total Score at Week 6 (fITT Population
Description: as for outcome 7
Time Frame: Baseline and Week 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Placebo | JNJ-42165279 25 mg
Number analyzed (Participants) | 72 | 69
Units on a Scale | -5.0 (6.95) | -5.6 (5.86)

9. Secondary Outcome: Double-blind Treatment Period: Change From Baseline in the HDRS17 Anxiety/Somatization Factor Total Score at Week 6 (eITT Population)
Description: The HDRS17 anxiety/somatization factor derived from Cleary and Guy's factor analysis of the HDRS17 scale, includes six items from the original 17-item version: psychic anxiety, somatic anxiety, gastrointestinal somatic symptoms, general somatic symptoms, hypochondriasis, and insight. Each of 6 items is rated by clinician on either a 3-point (0 to 2) or a 5-point (0 to 4) scale with rating of 0:absent, 1: doubtful to mild, 2: mild to moderate, 3: moderate to severe, and 4: very severe and is calculated as sum of 6 item scores ranging from 0 to 18, with higher scores indicating greater severity of symptoms for each item as well as total score.
Time Frame: Baseline and Week 6
Population: The eITT analysis set included all enrolled participants who were randomized into double blind treatment period, who were lead-in placebo non-responder, who received at least one dose of double-blind study medication (either placebo or JNJ-42165279) and had at least one post-baseline HDRS17 assessment in double-blind treatment period. Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | JNJ-42165279 25 mg
Number analyzed (Participants) | 47 | 47
Units on a scale | -2.1 (2.35) [lower limit 2.35] | -2.3 (1.55) [lower limit 1.55]

10. Secondary Outcome: Double-blind Treatment Period: Change From Baseline in the HDRS17 Anxiety/Somatization Factor Total Score at Week 6 (fITT Population)
Description: as for outcome 9
Time Frame: Baseline and Week 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Unit on a Scale
Arm/Group | Placebo | JNJ-42165279 25 mg
Number analyzed (Participants) | 72 | 69
Unit on a Scale | -1.7 (2.36) | -1.8 (1.69)

11. Secondary Outcome: Double-blind Treatment Period: Percentage of Participants With Greater Than or Equal to (>=) 30 Percent (%) Improvement on the HDRS17 Total Score at Week 6 (eITT Population)
Description: Percentage of participants who had >=30% improvement (responders) on HDRS17 total score at Week 6 were reported. HDRS17 is clinician-administered rating scale designed to assess severity of symptoms in participants diagnosed with depression. Each of 17 items is rated by clinician on either 3-point (0-2) or 5-point (0-4) scale with rating of 0: absent, 1: doubtful to mild, 2: mild to moderate, 3: moderate to severe, and 4: very severe. A total score (0 to 52) was calculated by adding scores of all 17 items. For each item as well as total score, higher score represents more severe condition.
Time Frame: Week 6
Population: as for outcome 9
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | JNJ-42165279 25 mg
Number analyzed (Participants) | 47 | 47
Percentage of participants | 51.1 | 55.3

12. Secondary Outcome: Double-blind Treatment Period: Percentage of Participants With >= 30 % Improvement on the HDRS17 Total Score at Week 6 (fITT Population)
Description: Percentage of participants who had >=30% improvement (responders) on HDRS17 total score at Week 6 was reported. HDRS17 is clinician-administered rating scale designed to assess severity of symptoms in participants diagnosed with depression. Each of 17 items is rated by clinician on either 3-point (0-2) or 5-point (0-4) scale with rating of 0: absent, 1: doubtful to mild, 2: mild to moderate, 3: moderate to severe, and 4: very severe. A total score (0 to 52) was calculated by adding scores of all 17 items. For each item as well as total score, higher score represents more severe condition.
Time Frame: Week 6
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | JNJ-42165279 25 mg
Number analyzed (Participants) | 72 | 69
Percentage of participants | 56.9 | 52.2

13. Secondary Outcome: Double-blind Treatment Period: Percentage of Participants With >= 50% Improvement in the HDRS17 Total Score at Week 6 (eITT Population)
Description: Percentage of participants who had >=50% improvement (responders) in HDRS17 total score at Week 6 were reported. HDRS17 is clinician-administered rating scale designed to assess severity of symptoms in participants diagnosed with depression. Each of 17 items is rated by clinician on either 3-point (0-2) or 5-point (0-4) scale with rating of 0: absent, 1: doubtful to mild, 2: mild to moderate, 3: moderate to severe, and 4: very severe. A total score (0 to 52) was calculated by adding scores of all 17 items. For each item as well as total score, higher score represents more severe condition.
Time Frame: Week 6
Population: The eITT analysis set included all enrolled participants who were randomized into double blind treatment period, who were lead-in placebo non-responder, who received at least one dose of double-blind study medication (either placebo or JNJ-42165279) and had at least one post-baseline HDRS17 assessment in DB treatment period. Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | JNJ-42165279 25 mg
Number analyzed (Participants) | 47 | 47
Percentage of participants | 27.7 | 21.3

14. Secondary Outcome: Double-blind Treatment Period: Percentage of Participants With >= 50% Improvement in the HDRS17 Total Score at Week 6 (fITT Population)
Description: as for outcome 13
Time Frame: Week 6
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | JNJ-42165279 25 mg
Number analyzed (Participants) | 72 | 69
Percentage of participants | 36.1 | 27.5

15. Secondary Outcome: Double-blind Treatment Period: Percentage of Participants With >= 30% Improvement on SIGH-A Total Score at Week 6 (eITT Population)
Description: The SIGH-A was included as a means to determine the frequency and severity of signs and symptoms of anxiety and determine both their influence on treatment and their responsiveness to treatment. The percentage of participants who had >= 30% improvement (responders) on SIGH-A total score at Week 6 was reported. The SIGH-A scale consists of 14 items with a score of 0 to 4, where 0=absent, 1=mild, 2=moderate, 3=severe, 4=incapacitating. The SIGH-A total score is calculated by summing the 14 item scores, and ranges from 0 to 56. For each individual item score and total score, higher scores indicate greater severity.
Time Frame: Week 6
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | JNJ-42165279 25 mg
Number analyzed (Participants) | 47 | 47
Percentage of participants | 48.9 | 51.1

16. Secondary Outcome: Double-blind Treatment Period: Percentage of Participants With >= 30% Improvement on SIGH-A Total Score at Week 6 (fITT Population)
Description: as for outcome 15
Time Frame: Week 6
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | JNJ-42165279 25 mg
Number analyzed (Participants) | 72 | 69
Percentage of participants | 52.8 | 52.2

17. Secondary Outcome: Double-blind Treatment Period: Percentage of Participants With >= 50% Improvement on SIGH-A Total Score at Week 6 (eITT Population)
Description: The SIGH-A was included as a means to determine the frequency and severity of signs and symptoms of anxiety and determine both their influence on treatment and their responsiveness to treatment. The percentage of participants who had >= 50% improvement (responders) on SIGH-A total score at Week 6 was reported. The SIGH-A scale consists of 14 items with a score of 0 to 4, where 0=absent, 1=mild, 2=moderate, 3=severe, 4=incapacitating. The SIGH-A total score is calculated by summing the 14 item scores, and ranges from 0 to 56. For each individual item score and total score, higher scores indicate greater severity.
Time Frame: Week 6
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | JNJ-42165279 25 mg
Number analyzed (Participants) | 47 | 47
Percentage of participants | 29.8 | 21.3

18. Secondary Outcome: Double-blind Treatment Period: Percentage of Participants With >= 50% Improvement on SIGH-A Total Score at Week 6 (fITT Population)
Description: as for outcome 17
Time Frame: Week 6
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | JNJ-42165279 25 mg
Number analyzed (Participants) | 72 | 69
Percentage of participants | 37.5 | 24.6

19. Secondary Outcome: Double-blind Treatment Period: Percentage of Participants With Remission as Assessed by HDRS17 Total Score Less Than or Equal to (<=) 7 at Week 6 (eITT Population)
Description: Percentage of participants with HDRS17 total score <= 7 were considered as remitters. HDRS17 is clinician-administered rating scale designed to assess severity of symptoms in participants with depression. Each of 17 items is rated by clinician on either 3-point(0-2) or 5-point(0-4) scale with rating of 0: absent, 1: doubtful to mild, 2: mild to moderate, 3: moderate to severe, and 4: very severe. A total score (0 to 52) was calculated by adding scores of all 17 items. For each item as well as total score, higher score represents more severe condition.
Time Frame: Week 6
Population: The eITT analysis set included all enrolled participants who were randomized into double-blind treatment period, who were lead-in placebo non-responder,who received at least one dose of double-blind study medication (either placebo or JNJ-42165279) and had at least one post-baseline HDRS17 assessment in double-blind treatment period. Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | JNJ-42165279 25 mg
Number analyzed (Participants) | 47 | 47
Percentage of participants | 14.9 | 8.5

20. Secondary Outcome: Double-blind Treatment Period: Percentage of Participants With Remission as Assessed by HDRS17 Total Score <= 7 at Week 6 (fITT Population)
Description: as for outcome 19
Time Frame: Week 6
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | JNJ-42165279 25 mg
Number analyzed (Participants) | 72 | 69
Percentage of participants | 33.3 | 21.7

21. Secondary Outcome: Double-blind Treatment Period: Percentage of Participants With a Clinical Global Impression Improvement (CGI-I) Score of Very Much Improved or Much Improved at Week 6 (eITT Population)
Description: The percentage of participants with a CGI-I score of very much improved or much improved at Week 6 was reported. CGI-I is a 7-point scale that required the clinician to assess how much the participant's illness had improved or worsened relative to a baseline state at the beginning of the intervention. The CGI-I is rated as: 1=very much improved; 2=much improved; 3=minimally improved; 4=no change; 5=minimally worse; 6=much worse; 7=very much worse. For each individual item score and total score, higher scores indicate greater severity.
Time Frame: Week 6
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | JNJ-42165279 25 mg
Number analyzed (Participants) | 47 | 47
Percentage of participants | 57.4 | 55.3

22. Secondary Outcome: Double-blind Treatment Period: Percentage of Participants With a Clinical Global Impression Improvement (CGI-I) Score of Very Much Improved or Much Improved at Week 6 (fITT Population)
Description: as for outcome 21
Time Frame: Week 6
Population: as for outcome 6
Measure: Number; unit: Percentage of participate
Arm/Group | Placebo | JNJ-42165279 25 mg
Number analyzed (Participants) | 72 | 69
Percentage of participate | 65.3 | 65.2

23. Secondary Outcome: Maximum Plasma Concentration (Cmax) of JNJ-42165279
Description: Cmax is defined as maximum plasma concentration of JNJ-42165279. The data was pooled across visits at different timepoints to calculate Cmax.
Time Frame: Pre-dose, 2 to 4 hours post-dose on Days 14, 35, 63, and 77
Population: The Pharmacokinetic analysis set included all participants who received at least 1 dose of JNJ-42165279 and with measurable JNJ-42165279 concentrations in plasma. Here "n (number analyzed)" is defined as number of participants analyzed for specified categories.
Measure: Mean (90% Confidence Interval); unit: Nanograms/milliliter (ng/mL)
Arm/Group | JNJ-42165279 25 mg
Number analyzed (Participants) | 77
Nanograms/milliliter (ng/mL)
  Male: number analyzed (Participants) | 24
  Male | 217.7 [178.4 to 281.7]
  Female: number analyzed (Participants) | 53
  Female | 229.3 [142.9 to 337.7]

24. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Zero to Dosing Intervals (AUC[0-tau]) of JNJ-42165279
Description: AUC(0-tau) is defined as area under the plasma concentration-time curve from 0 to t hours post dosing (time t is the dosing interval). The data was pooled across visits at different timepoints to calculate AUC(0-tau).
Time Frame: Pre-dose, 2 to 4 hours post-dose on Days 14, 35, 63, and 77
Population: The Pharmacokinetic analysis set included all participants who received at least 1 dose of JNJ-42165279 and with measurable JNJ-42165279 concentrations in plasma. Here "n (number analyzed)" is defined as number of participants analyzed for specified category.
Measure: Mean (90% Confidence Interval); unit: Nanograms*hour/milliliter (ng*h/mL)
Arm/Group | JNJ-42165279 25 mg
Number analyzed (Participants) | 77
Nanograms*hour/milliliter (ng*h/mL)
  Male: number analyzed (Participants) | 24
  Male | 2159 [1353 to 3385]
  Female: number analyzed (Participants) | 53
  Female | 2432 [1137 to 4288]

25. Secondary Outcome: Time to Reach the Maximum Plasma Concentration (Tmax) of JNJ-42165279
Description: Tmax is defined as time to reach the maximum plasma concentration of JNJ-42165279. The data was pooled across visits at different timepoints to calculate Tmax.
Time Frame: Pre-dose, 2 to 4 hours post-dose on Days 14, 35, 63, and 77
Population: The Pharmacokinetic analysis set included all participants who received at least 1 dose of JNJ-42165279 and with measurable JNJ-42165279 concentrations in plasma. Sparse samples was collected between 2 hours and 4 hours. It was not possible to accurately determine Tmax as Cmax is expected to be around 1 hour post-dose.
Measure: Median (Full Range); unit: Hours
Arm/Group | JNJ-42165279 25 mg
Number analyzed (Participants) | 77
Hours | NA [NA to NA] — With the sparse sampling collected between 2 and 4 hours it was not possible to accurately determine Tmax as Cmax is expected to be around 1h post-dose.

ADVERSE EVENTS:
Time Frame: Up to Week 18
Description: Safety analysis set included all randomized participants who received at least 1 dose of study drug.
Groups:
- Double-blind (DB) Lead-in Period: Placebo: All participants received matching placebo tablets orally once daily (qd) during the double blind lead-in period.
- DB Treatment + Withdrawal Period: Placebo: All participants received matching placebo tablets orally qd during the double blind lead-in period. Participants were then assessed for response according to criteria based on reduction from lead-in baseline in Hamilton depression rating scale (HDRS17) and continued to receive adjunctive matching placebo tablets orally qd for 6 weeks during the double-blind treatment period. Participants who completed the double-blind treatment period prior to Week 11 entered the withdrawal period and were treated with placebo for the remaining time of the treatment phase of the study, which varied depending on the duration of the placebo lead-in for the specific participant.
- DB Treatment + Withdrawal Period: JNJ-42165279 25 mg: Participants receiving matching placebo tablets during the double blind lead-in period were randomized to receive JNJ-42165279 25 milligrams (mg) tablets orally qd for 6 weeks during the double-blind treatment period. Participants who completed the double-blind treatment period prior to Week 11 entered the withdrawal period and were treated with placebo for the remaining time of the treatment phase of the study, which varied depending on the duration of the placebo lead-in for the specific participant.
Arm/Group | Double-blind (DB) Lead-in Period: Placebo | DB Treatment + Withdrawal Period: Placebo | DB Treatment + Withdrawal Period: JNJ-42165279 25 mg
All-Cause Mortality (participants affected / at risk) | 0/160 | 0/76 | 0/77
Serious Adverse Events (participants affected / at risk) | 2/160 | 1/76 | 1/77
Other Adverse Events (participants affected / at risk) | 16/160 | 4/76 | 3/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind (DB) Lead-in Period: Placebo (N=160) | DB Treatment + Withdrawal Period: Placebo (N=76) | DB Treatment + Withdrawal Period: JNJ-42165279 25 mg (N=77)
Gastroenteritis (Infections and infestations) | 1 | 1 | 0
Foot Deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind (DB) Lead-in Period: Placebo (N=160) | DB Treatment + Withdrawal Period: Placebo (N=76) | DB Treatment + Withdrawal Period: JNJ-42165279 25 mg (N=77)
Headache (Nervous system disorders) | 16 | 4 | 3

LIMITATIONS AND CAVEATS:
The relationship of plasma anandamide and trough drug concentrations observed suggest that few participants had substantial recovery of fatty acid amide hydrolase activity between doses. Higher doses or exposures could have resulted in greater effects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2017-10-24): https://cdn.clinicaltrials.gov/large-docs/92/NCT02498392/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-14): https://cdn.clinicaltrials.gov/large-docs/92/NCT02498392/SAP_001.pdf